CLINICAL TRIAL: NCT05538182
Title: Zimbabwe Eyecare And Learning: Formative Research on Hyperopia and Educational Outcomes in Primary School Children in Mashonaland Central Province of Zimbabwe
Brief Title: Zimbabwe Eyecare And Learning(ZEAL):Formative Research on Hyperopia and Educational Outcomes in Primary School Children
Acronym: ZEAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: L.V. Prasad Eye Institute (Other); University of Zimbabwe (Other); University of Ulster (Other); New England College of Optometry (Other); Peek Vision (Unknown); Zimbabwe Optometric Association (Unknown); Clearly (Other); Christian Blind Mission (Unknown)
Responsible Party: Principal Investigator, Nathan Congdon, Professor, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHLS 22_63
Record Dates: First submitted 2022-09-09; First posted 2022-09-13 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Hyperopia; Long Sight
Keywords: Refractive error; Spectacle correction; Eyeglasses; Learning; School children
MeSH Terms: conditions — Hyperopia; Refractive Errors | interventions — Eyeglasses

STUDY DESIGN:
Intervention Model Description: Children in Grade 2 and 4 at 16 randomly-selected primary schools in Mashonaland Central province of Zimbabwe will receive free glasses as described in the protocol.
Who Masked: Outcomes Assessor
Masking Description: For the following objectives, all tests will be conducted by trained researchers who will be masked to the hyperopia status of the children:
  1. Prevalence of moderate to high hyperopia (>+2.00D in the more hyperopic meridian, in the more hyperopic eye, using cycloplegic autorefraction).
  2. The diagnostic accuracy of four screening tools for detecting hyperopia compared to the gold standard of cycloplegic refraction.
  3. The cross-sectional association between uncorrected moderate to high hyperopia and baseline reading levels (using the Happy Readers V4 tool). We will compare the results to age-, gender-and school-matched emmetropic children.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spectacles (Experimental): Based on the refraction results, spectacles will be prescribed at the baseline visit and worn throughout the study. Study participants with newly diagnosed hyperopia at baseline will undergo a reading assessment and near visual acuity check over six months, compared to age-, gender- and school-matched emmetropic controls.
  Spectacle compliance will be observed among newly diagnosed hyperopic and newly diagnosed myopic school children in Grades 2 and 4 primary school children, from Mashonaland Central province of Zimbabwe, at six weeks and 14 weeks from spectacle acquisition.
  Interventions: Device: Spectacles
- No treatment (No Intervention): Age-, gender- and school-matched emmetropic controls will undergo a reading assessment at baseline and at six months.

INTERVENTIONS:
Device: Spectacles — Based on the refraction results, study participants diagnosed with refractive error will be dispensed two free pairs of distance spectacles.
  Arms: Spectacles

SUMMARY:
The purpose of this study is to determine whether uncorrected or corrected long-sightedness (hyperopia) has an impact on reading skills, in Grade 2 or Grade 4 school-aged children from Mashonaland Central province of Zimbabwe, compared to age-, gender- and school-matched children with no refractive error (emmetropia), measured by the Happy Readers V4 reading tool over six months.

DETAILED DESCRIPTION:
Trials in Asia have shown that correction of myopia (close-sightedness) in children has improved educational performance with an effect size larger than for any other school-based health intervention. Myopia prevalence which is, generally inversely associated with the prevalence of hyperopia, appears low in African children. Globally, uncorrected hyperopia (long-sightedness) has a higher prevalence and is present in 12-26% of children, depending on location and age, but the impact of its correction on educational outcomes is not well understood. All-age prevalence of hyperopia is higher in Africa than in any other global region. Despite the traditional view that moderate hyperopia is generally benign, emerging evidence suggests that even moderate uncorrected hyperopia is associated with reduced near function, poorer educational outcomes and lower reading scores. A recent trial in the USA showed that providing refractive correction improved reading scores but did not distinguish between myopia and hyperopia. Another trial in the USA found only small benefits from refractive correction in 1- to 2-year-olds. However, no trial to date has studied the educational impact of hyperopic correction in school-aged children with +2.00 Dioptres (D) or more of hyperopia.

While the gold standard for detecting hyperopia in children during vision examinations requires cycloplegic eye drops to temporarily inhibit accommodation (focusing effort to see near objects), using these eye drops requires trained providers and clinical supervision. It is not typically feasible in vision screening settings. The Vision in Preschoolers study showed that two autorefractors (Retinomax, SureSight) and non-cycloplegic retinoscopy had high discriminatory power to detect young children with hyperopia. However, non-cycloplegic retinoscopy requires trained providers, SureSight is no longer commercially available, and the Retinomax is cost-prohibitive for many screening programs. This limits the availability of hyperopia prevalence data in African children, though, as noted above, available evidence suggests high rates. Most screening programmes use 6/12 as an optimal cut-off value for distance vision. However, studies have reported that measuring distance vision alone is ineffective in detecting hyperopia. Literacy rates remain particularly low among primary school children in sub-Saharan Africa compared to other regions. The challenges and importance of maximising children's early learning, and the potentially important role of vision correction, are not well-understood in this setting. However, these initiatives have focused on myopia, not hyperopia.

Study plan: 2000 study participants (1000: Grade 2, 1000: Grade 4) will be recruited from primary schools selected by the Ministry of Primary and Secondary Education (MoPSE) in Mashonaland Central province in Zimbabwe.

Study design:

Objectives 1, 2 and 3 use a cross-sectional study design to assess the following:

1. To assess the prevalence of moderate to high hyperopia (≥ +2.00D) among primary school children in Grades 2 and 4 from Mashonaland Central province in Zimbabwe.
2. To accurately detect moderate to high hyperopia (≥ +2.00D) using four screening tests compared to the gold-standard cycloplegic refraction.
3. To study the association between uncorrected and corrected moderate to high hyperopia (≥ +2.00D) and baseline reading levels.

   Objectives 4 and 5 use a longitudinal intervention design to assess the following:
4. To compare near visual acuity and reading levels at baseline and at six months between moderate to high hyperopic (≥ +2.00D) children compared to age-, gender-, and school-matched controls with no vision problems.
5. To compare spectacle compliance among newly diagnosed hyperopic and newly diagnosed myopic (short-sighted) school children at six weeks and 14 weeks.

ELIGIBILITY:
Inclusion criteria for the cross-sectional assessment of hyperopia prevalence and diagnostic tool development evaluation:

* Grades 2 or 4 from the list of selected primary schools by the Ministry of Primary and Secondary Education (MoPSE)

Inclusion criteria for the baseline and longitudinal assessment of reading performance

Primary school children will be eligible to participate in the 'reading assessment' if they fulfil the following criteria:

Hyperopic cohort:

* In Grade 2 or 4 from the list of selected schools by the MoPSE.
* Presence of moderate to high hyperopia, defined as ≥ +2.00D in the more hyperopic meridian, in the more hyperopic eye, using cycloplegic autorefraction with an average of three consecutive readings taken.

Emmetropic cohort:

* In Grade 2 or 4 from the list of selected schools by the MoPSE.
* Meets criteria for visually normal (unaided distance visual acuity 6/6 monocular and near visual acuity N5), based on an absence of significant refractive error.
* Presence of emmetropia, defined as < +1.00D to >-0.50 Dioptre in the more hyperopic meridian, in both eyes using cycloplegic autorefraction with an average of three consecutive readings taken to record the refractive status.

Newly diagnosed hyperopic and newly diagnosed myopic children will be eligible to participate in the 'spectacle compliance' assessment if they fulfil the following criteria:

Hyperopic cohort:

* Presence of hyperopia, defined as ≥ +2.00D in the more hyperopic meridian, in the more hyperopic eye by cycloplegic autorefraction.

Myopic cohort:

* Presence of myopia, defined as <-0.50D in the more hyperopic meridian, in either eye by cycloplegic autorefraction.

Exclusion criteria for the baseline and longitudinal assessment of reading performance and spectacle compliance.

Children in either cohort will be ineligible if they have:

* History of systemic disease or ocular disease and/or medications known to have an impact on accommodation.
* History of previous spectacle wear

Children in the hyperopic cohort will be ineligible if they have:

* Vision limitation in either eye for reasons other than hyperopia (including amblyopia defined as <6/12 in the better eye).

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1883 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Prevalence of moderate to high hyperopia (≥ +2.00D) | Measured at baseline
  The metric or method of measurement to be used:The Average of three readings(in dioptre)using cycloplegic autorefraction for each eye. Higher dioptre indicates high hyperopia
Binocular near visual acuity | Measured at baseline
  The metric or method of measurement to be used: Logarithm of Minimum Angle of Resolution(LogMAR) measured using the laser-etched near vision chart with Lea symbols at 12.5 cm.
Accommodative response | Measured at baseline
  The metric or method of measurement to be used: binocular distance autorefraction measured at 3 metres and monocular near refraction measured at 25cm using the Quick See autorefractor.
Presence of eye conditions | Measured at baseline
  The metric or method of measurement to be used: assessing the overall appearance of the fundus reflex in both eyes(Bruckner Reflex Test) as an indicator of the prevalence of refractive error using the Arclight ophthalmoscope. This will be a binary outcome of Yes or No.
Stereoacuity | Measured at baseline
  The metric or method of measurement to be used: measured in seconds of arc using the Preschool Assessment of Stereopsis with a Smile (PASS) 3+ stereoacuity test (scores: 480, 240, 120, 60, 40 and 30). Seconds of arc refers to the visual angle being measured to determine depth perception. Lower scores indicate better stereoacuity.
  Highest possible score: 480 Lowest possible score: 30
Improvement in near visual acuity on prescribing hyperopic spectacle correction | Measured at baseline,2 weeks and 24 weeks after baseline
  The metric or method of measurement to be used: measured in M-unit using a conventional near vision chart with Lea symbols at 40cm.
Change of reading scores 6 months post hyperopia spectacle correction | Measured at baseline and at month -6
  The metric or method of measurement to be used: Reading scores measured using the Happy Readers V4 reading test.
  Best possible score: Improvement from baseline Worst possible score: No change from baseline
Observed spectacle wear | Measured at week 6 and week 14 from baseline
  The metric or method of measurement to be used: proportion of children prescribed with spectacles, wearing them during unannounced direct observation

CONTACTS AND LOCATIONS:
Overall Officials: Nathan G Congdon, MD, MPH, Principal Investigator — Queen's University, Belfast; Rohit C Khanna, MPH, Principal Investigator — L.V. Prasad Eye Institute; Lynett E Masiwa, MSc, Principal Investigator — University of Zimbabwe; Rangarirai Masanganise, Principal Investigator — University of Zimbabwe
Locations (1):
- The University of Zimbabwe, Faculty of Medicine and Healthcare Sciences, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
All Individual Participant Data (IPD) will be stored in an anonymised format. The IPD that includes personally identifiable information will be deleted when the data collection process is complete and before the initiation of data analysis.
  Only de-identified data will be shared with all the researchers for analysis. The primary analysis will be conducted on all outcome data obtained from all enrolled participants as randomised.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: All deidentified IPD will be available from June 2022 (anticipated Trial start date) to December 2032 (inclusive of analysis, publication and archival).
Access Criteria: Following publication of the primary outcomes there may be scope to conduct additional analyses on the data collected. In such instances formal requests for data will need to be made in writing to the Chief Investigator, who will discuss this with the Sponsor. The study will comply with the good practice principles for sharing individual participant data from publicly funded clinical trials and data sharing will be undertaken in accordance with the required regulatory requirements.

REFERENCES:
- [Background] Ma X, Zhou Z, Yi H, Pang X, Shi Y, Chen Q, Meltzer ME, le Cessie S, He M, Rozelle S, Liu Y, Congdon N. Effect of providing free glasses on children's educational outcomes in China: cluster randomized controlled trial. BMJ. 2014 Sep 23;349:g5740. doi: 10.1136/bmj.g5740. PMID 25249453
- [Background] Ma Y, Congdon N, Shi Y, Hogg R, Medina A, Boswell M, Rozelle S, Iyer M. Effect of a Local Vision Care Center on Eyeglasses Use and School Performance in Rural China: A Cluster Randomized Clinical Trial. JAMA Ophthalmol. 2018 Jul 1;136(7):731-737. doi: 10.1001/jamaophthalmol.2018.1329. PMID 29801081
- [Background] Glewwe P, West KL, Lee J. The Impact of Providing Vision Screening and Free Eyeglasses on Academic Outcomes: Evidence from a Randomized Trial in Title I Elementary Schools in Florida. J Policy Anal Manage. 2018;37(2):265-300. doi: 10.1002/pam.22043. PMID 29693366
- [Background] Narayanasamy S, Vincent SJ, Sampson GP, Wood JM. Impact of simulated hyperopia on academic-related performance in children. Optom Vis Sci. 2015 Feb;92(2):227-36. doi: 10.1097/OPX.0000000000000467. PMID 25525890
- [Background] Naidoo KS, Raghunandan A, Mashige KP, Govender P, Holden BA, Pokharel GP, Ellwein LB. Refractive error and visual impairment in African children in South Africa. Invest Ophthalmol Vis Sci. 2003 Sep;44(9):3764-70. doi: 10.1167/iovs.03-0283. PMID 12939289
- [Background] O'Donoghue L, McClelland JF, Logan NS, Rudnicka AR, Owen CG, Saunders KJ. Refractive error and visual impairment in school children in Northern Ireland. Br J Ophthalmol. 2010 Sep;94(9):1155-9. doi: 10.1136/bjo.2009.176040. Epub 2010 May 21. PMID 20494909
- [Background] French AN, O'Donoghue L, Morgan IG, Saunders KJ, Mitchell P, Rose KA. Comparison of refraction and ocular biometry in European Caucasian children living in Northern Ireland and Sydney, Australia. Invest Ophthalmol Vis Sci. 2012 Jun 26;53(7):4021-31. doi: 10.1167/iovs.12-9556. PMID 22562516
- [Background] Hashemi H, Fotouhi A, Yekta A, Pakzad R, Ostadimoghaddam H, Khabazkhoob M. Global and regional estimates of prevalence of refractive errors: Systematic review and meta-analysis. J Curr Ophthalmol. 2017 Sep 27;30(1):3-22. doi: 10.1016/j.joco.2017.08.009. eCollection 2018 Mar. PMID 29564404
- [Background] Babinsky E, Candy TR. Why do only some hyperopes become strabismic? Invest Ophthalmol Vis Sci. 2013 Jul 24;54(7):4941-55. doi: 10.1167/iovs.12-10670. PMID 23883788
- [Background] VIP-HIP Study Group; Kulp MT, Ciner E, Maguire M, Moore B, Pentimonti J, Pistilli M, Cyert L, Candy TR, Quinn G, Ying GS. Uncorrected Hyperopia and Preschool Early Literacy: Results of the Vision in Preschoolers-Hyperopia in Preschoolers (VIP-HIP) Study. Ophthalmology. 2016 Apr;123(4):681-9. doi: 10.1016/j.ophtha.2015.11.023. Epub 2016 Jan 27. PMID 26826748
- [Background] Shankar S, Evans MA, Bobier WR. Hyperopia and emergent literacy of young children: pilot study. Optom Vis Sci. 2007 Nov;84(11):1031-8. doi: 10.1097/OPX.0b013e318157a67a. PMID 18043422
- [Background] Rosner J, Rosner J. The relationship between moderate hyperopia and academic achievement: how much plus is enough? J Am Optom Assoc. 1997 Oct;68(10):648-50. PMID 9354056
- [Background] Williams WR, Latif AH, Hannington L, Watkins DR. Hyperopia and educational attainment in a primary school cohort. Arch Dis Child. 2005 Feb;90(2):150-3. doi: 10.1136/adc.2003.046755. PMID 15665167
- [Background] Atkinson J, Braddick O, Nardini M, Anker S. Infant hyperopia: detection, distribution, changes and correlates-outcomes from the cambridge infant screening programs. Optom Vis Sci. 2007 Feb;84(2):84-96. doi: 10.1097/OPX.0b013e318031b69a. PMID 17299337
- [Background] Glewwe P, Park A, Zhao M. A better vision for development: Eyeglasses and academic performance in rural primary schools in China. J Dev Econ. 2016;122:170-82.
- [Background] White SLJ, Wood JM, Black AA, Hopkins S. Vision screening outcomes of Grade 3 children in Australia: Differences in academic achievement. Int J Educ Res. 2017;83:154-9.
- [Background] Slavin RE, Collins ME, Repka MX, Friedman DS, Mudie LI, Owoeye JO, et al. In Plain Sight: Reading Outcomes of Providing Eyeglasses to Disadvantaged Children. J Educ Stud Placed Risk. 2018;23(3):250-8.